CLINICAL TRIAL: NCT05141032
Title: Prospective Registry of Endoscopic Resection Procedures Performed With the Assistance of a Novel Rigidizing Overtube
Brief Title: Pathfinder Registry
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Salmaan Azam Jawaid, MD, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-49475
Record Dates: First submitted 2021-11-17; First posted 2021-12-02 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Polyps
Keywords: Endoscopic Submucosal Dissection
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Research Subject: Only one group will be made which will contain all subjects recruited into research study.
  Interventions: Procedure: Endoscopic Submucosal Dissection with Pathfinder/Overtube device

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection with Pathfinder/Overtube device — Removal of gastrointestinal polyps via ESD

SUMMARY:
This study collects information regarding your procedure. No changes will be done to your procedure and you are asked to consent for the use of your data in our database. You are being asked to be in this research study because you have a gastrointestinal lesion that needs to be removed. We remove these lesions endoscopically as part of the standard of care at Baylor St. Luke Medical Center, and we will be using a FDA approved device known as the Pathfinder Rigidization Overtube to assist with the removal of the polyp. This study is important because this is a relatively new procedure; although it is a part of your standard of care it is not done in many hospitals. We would like to document the outcomes and results of such procedures to continuously improve our standard of care.

DETAILED DESCRIPTION:
All patients will receive standard medical care and no experimental interventions will be performed. The Pathfinder Overtube is already being used to assist in polyp removal at our center and many other centers, thus the device itself is not experimental. All patients scheduled to undergo ESD or EMR for colonic lesions at the Baylor St Luke's Medical Center as medically indicated and standard of care will be considered for the study. Patients for whom ESD or EMR is considered as part of their standard medical care will be offered to participate in this study. The patients involvement in the study does not preclude the use of the Pathfinder Overtube. If the patient does not agree to participate, outcomes related to the use of the Pathfinder Overtube or personal information will not be recorded. The Pathfinder Overtube will still be used to assist in the removal of polyps as deemed appropriate by the endoscopist. The physician performing the procedure will also discuss the study with the subjects and ask them to sign a consent. If the patient agrees to participate, he or she will be given the informed consent form and allowed enough time to read it. Opportunity to ask questions will be provided.

Data collection: After obtaining the informed consent, the following information will be collected from the subject's chart regarding the procedure:

1- Demographic information related to the study participants (age, sex, race, MRN etc.) 2- Comorbid conditions of the study participant (prior history of hysterectomy, or other abdominal surgeries) 3- Total en bloc resection rate. 4- Total E0 resection rate. 5- Total length of procedure time. 6- Total number of polyps detected, 7- Stabilization within the gastrointestinal lumen 8- Complications within 1 week after the procedure (perforation, bleeding) Equipment and techniques: All procedures will be performed with the Pathfinder Overtube (already FDA approved for use within the gastrointestinal lumen) and 19-inch high-definition monitor (OEV 191H; OlympusAmerica Inc.).

If the patient agrees to participate, he or she will sign the consent form and a copy will be provided. Data will be prospectively recorded according to the data collection form. ESD or EMR with Pathfinder Overtube will be performed as medically indicated. Follow-up will be carried out as medically indicated and no additional studies or clinic visits will be needed specifically for the purpose of this study. Data collection will last approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-80 years) Any gastrointestinal polyp that has been deemed appropriate for endoscopic removal.

Exclusion Criteria:

* Pregnant patients
* Prisoners
* Unable to sign consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have been found to have duodenal or colon polyps will be identified as potential suitable subjects.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Technical success | Day 1
  Defined by the completion of endoscopic submucosal dissection (ESD) or endoscopic mucosal resection (EMR) procedure while utilizing the Rigidization Overtube.
Procedure feasibility | Day 1
  Defined by the ability of endoscopist to reach lesion of interest while using the Rigidization Overtube for ESD/EMR procedures and complete entire procedure with device. This will be assessed as a rate (percentage).

SECONDARY OUTCOMES:
En bloc resection rate | Day 1
  En bloc resection rate using the Rigidization Overtube.
R0 resection rate | 3-5 days
  To evaluate the R0 resection rates by assessing lesion margins while using the Rigidization Overtube.
Procedure time | Day 1
  Determine overall procedure times using the Rigidizing Overtube.

OTHER OUTCOMES:
Complications | 2 weeks
  Issues arising immediately or post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States